CLINICAL TRIAL: NCT06293300
Title: Understanding and Treating TBI Associated Photophobia With Botulinum Toxin Type A and Its Impact on Visual Function
Brief Title: Understanding and Treating Traumatic Brain Injury (TBI) Associated Photophobia With Botulinum Toxin Type A (BoNT-A)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anat Galor, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231056; HT94252310608 (Other Grant/Funding Number: Department of Defense Awarding Office: U.S. Army Medical Research Acquisition Activity (USAMRAA))
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BoNT-A Group (Experimental): Participants will receive BoNT-A intervention for up to 6 months.
  Interventions: Drug: BoNT A

INTERVENTIONS:
Drug: BoNT A — Participants with TBI-associated photophobia will come one time in person to the clinic and receive 35 Units of BoNT-A injected in 7 forehead sites (0.1 cc in each location).

SUMMARY:
The purpose of this research is to understand and treat Traumatic Brain Injury (TBI) associated photophobia (light sensitivity) and its impact on visual function.

ELIGIBILITY:
Inclusion Criteria:

* Recruit and enroll male and female subjects, civilians and veterans (1:1 mix anticipated, i.e., n = 25 from each group) of all races and ethnicities.
* ≥18 years of age who are able to consent.
* Report chronic photophobia (Numerical Rating Scale ≥4 on a 0-10 scale, photophobia present ≥6 months) with a remote history of TBI (>1 year).
* Inclusion into the study with regard to TBI status will be based on the Department of Defense Standard Surveillance Case Definition for TBI Adapted for Armed Forces Health Surveillance Division (AFHSB) Use. This can include one hospitalization or outpatient medical encounter with documented International Classification of Diseases (ICD9/ICD10) codes as identified within the Surveillance Case Definition.
* Subjects must also have been on a stable medication regimen for the past 3 months and must be naïve to BoNT-A treatment for orofacial conditions.
* English as primary language (by self-report).

Exclusion Criteria:

* Individuals with ocular diseases that may confound photophobia, such as glaucoma, corneal and conjunctival scarring, corneal edema, uveitis, iris transillumination defects, retinal degeneration, etc.
* Patients who are participating in another study with an investigational drug within one month prior to screening.
* Pregnant individuals. Pregnant subjects will not be scanned in the functional Magnetic Resonance Imaging (fMRI). Although there are no known risks associated with MRI during pregnancy, according to facility policy, University of Miami will not scan someone that is pregnant. Therefore, all women of childbearing potential (menstruating or >12 years old) must complete a for stating that are not pregnant within 24 hours of each MRI scan.
* Individuals with contraindications to fMRI scanning (e.g. metal implants, pacemaker) will not be offered inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in photophobia measured by Numerical Rating Scale | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  The change in numerical rating of average photophobia during the past week, ranging from 0 (for "no ocular pain") to 10 ("the most intense ocular pain imaginable").
Change in visual photosensitivity thresholds (VPT) measured Ocular Photosensitivity Analyzer (OPA) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  The change in the OPA visual photosensitivity thresholds, ranging from 0 to 4.51 log lux, with a lower VPT indicating less tolerance to light or increased light sensitivity.

SECONDARY OUTCOMES:
Change in severity of visual photosensitivity symptoms measured by Visual Light Sensitivity Questionnaire-8 (VLSQ-8) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  Total score ranging from 8 to 40, with a higher score indicating more visual photosensitivity symptom severity.
Change in severity of neuropathic ocular pain symptoms measured by Neuropathic Pain Symptom Inventory Questionnaire, modified for the Eye (NPSI-Eye). | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  Total score ranging from 0 to 100, with higher scores reflecting greater neuropathic ocular pain symptom severity.
Change in visual function related to activities of daily living measured by Visual Function Questionnaire-25 (VFQ-25) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  Total score ranging from 0 to 100, with higher scores indicating better quality of life.
Change in migraine symptom severity score measured by in Migraine Symptom Severity Score (MSSS) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  Total score ranging from 0 to 21, with higher scores indicating greater migraine severity.
Change in impact of headaches on daily life measured by Headache Impact Test (HIT)-6 | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  Total score ranging from 36 to 78, with higher scores indicating greater impact of headaches have on a person's ability to function on the job, at school, at home and in social situations.
Change in dry eye symptoms measured by the Dry Eye Questionnaire 5 (DEQ 5) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  Total score ranging from 0 to 22, with higher scores indicating more dry eye symptoms.
Change in ocular surface disease index measured by the Ocular Surface Disease Index (OSDI) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  Total score ranging from 0 to 100, will be administered to assess dry eye symptoms, with higher scores indicating more dry eye symptoms and impact on daily activities.
Change in pain intensity rating of aftersensations (AS) to repeated heat stimulation on the forehead measure by quantitative sensory testing (QST) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  QST methodology will be used to measure the severity of painful sensations that remain present 15 seconds after presentation of 10 one-second presentations (each separated by one second) of a noxious stimulus to the skin of the forehead. Ratings of the "intensity of pain" on a 0 to 100 numerical rating scale (0 = "no pain"; 100 = "most intense pain imaginable") will be recorded for these aftersensations.
Change in temporal summation (TS) of heat pain on the forehead measure by quantitative sensory testing (QST) | Baseline, 6-weeks post-intervention, and 12-weeks post-intervention.
  QST methodology will be used to measure the increase in pain intensity ratings that occur when repeated noxious stimuli are presented in rapid succession (i.e., temporal summation; TS). Ratings of the "intensity of pain" on a 0 to 100 numerical rating scale (0 = "no pain"; 100 = "most intense pain imaginable"). TS at each study time point will be determined by subtracting the rating of pain intensity at its peak during the rapid train of one-second noxious heat stimuli from the rating of pain intensity after a single one-second heat stimulus of the same temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Anat Galor, MD/MSPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No